CLINICAL TRIAL: NCT05041049
Title: Virtual Simulation Versus High-Fidelity Mannequin Simulation to Train Anesthesia Residents
Brief Title: Virtual Simulation Versus High-Fidelity Mannequin Simulation
Status: Approved for marketing | Type: Expanded Access
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Gianluca Bertolizio, Associate Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: 2021-7663
Record Dates: First submitted 2021-09-02; First posted 2021-09-10 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Comparing Visual Reality to High-fidelity Mannequin Stimulation

INTERVENTIONS:
Device: Comparing Visual Reality to High-fidelity mannequin Stimulation — This is a prospective, randomized, non-inferiority study. VR will be compared to HFS, which will be considered the a priori gold standard for residents simulation training.
  The study will be divided into two phases. In the pre-test phase, participants will be randomly allocated to receive either a VR or HFS scenario (scenario 1, see below). In the post-test phase, all participants (regardless the initial grouping) will undergo a HFS scenario (scenario 2, see below).
  All scenarios have been chosen from critical events published by the Society of Pediatric Anesthesia48 and adult sources49.
  The study will be conducted at the McGill University Health Center - Research Institute (MUHC-RI).
  Other Names: Comparing VR to HFS; To assess whether VR is as effective as mannequin-based HFS in anesthesia resident training.

SUMMARY:
Background. Despite remarkable progress, pediatric anesthesia-related mortality remains 2 to 30 times higher than in adults. Non-technical skills rather than a lack of expertise were identified to be the main cause of errors in medicine, particularly in emergency situations. As a consequence, interactive computer-based sessions and high-fidelity simulation have been progressively integrated into pediatric training programs. The setup of a suitable simulation center, however, is expensive and requires space, logistical support and manpower. Virtual reality (VR) is a technological innovation that has been increasingly integrated into clinical practice and medical training. Comparing to the mannequin-based simulation, theoretical advantages of VR are the inherent highly immersive quality, the independent participation with no need of other participants, the ease of multiple repetitions, the lack of time or space constrains, and the reduced costs. Non-technical and operational skills appear to improve significantly after VR training. To date, information on the efficacy of VR in the anesthesia training are limited.

Objectives. The primary aim will be to compare the improvement of non-technical skills after one simulation session between VR and high-fidelity mannequin simulation (HFS). Secondary aims will be to compare the overall anesthesia resident non-technical skills performance between VR and HFS, and to determine confidence in the simulation training of each participant.

Methods. This is a prospective, randomized, non-inferiority study. Eighteen residents in anesthesia (R1-R5) will be enrolled. Participants of each year will be randomly allocated to be involved in either a VR or a HFS training. The scenario will be the same for both VR and HFS groups. Within two weeks after the training session, all participants will undergo a different, mannequin-based HFS scenario.

After each simulation, resident performance will be assessed using the Anaesthetists' Non-Technical Skills scale and the Ottawa Crisis Resource Management Global Rating Scale. Evaluators will also perform a summary evaluation with the Managing Emergencies in Pediatric Anesthesia Global Rating Scale.

Resident's satisfaction will be measured with a post-assessment trainee survey scale.

Significance. Should the virtual reality demonstrate to be as efficient as mannequin-based simulation, it will be integrated into the residency curriculum and used for resident training and medical education in institutions that have limited access to a simulation center.

DETAILED DESCRIPTION:
Background. Despite remarkable progress, pediatric anesthesia-related mortality remains 2 to 30 times higher than in adults. Non-technical skills rather than a lack of expertise were identified to be the main cause of errors in medicine, particularly in emergency situations. As a consequence, interactive computer-based sessions and high-fidelity simulation have been progressively integrated into pediatric training programs. The setup of a suitable simulation center, however, is expensive and requires space, logistical support and manpower. Virtual reality (VR) is a technological innovation that has been increasingly integrated into clinical practice and medical training. Comparing to the mannequin-based simulation, theoretical advantages of VR are the inherent highly immersive quality, the independent participation with no need of other participants, the ease of multiple repetitions, the lack of time or space constrains, and the reduced costs. Non-technical and operational skills appear to improve significantly after VR training. To date, information on the efficacy of VR in the anesthesia training are limited.

Objectives. The primary aim will be to compare the improvement of non-technical skills after one simulation session between VR and high-fidelity mannequin simulation (HFS). Secondary aims will be to compare the overall anesthesia resident non-technical skills performance between VR and HFS, and to determine confidence in the simulation training of each participant.

Methods. This is a prospective, randomized, non-inferiority study. Twenty residents in anesthesia (R1-R5) will be enrolled. Participants of each year will be randomly allocated to be involved in either a VR or a HFS training. The scenario will be the same for both VR and HFS groups. Within three weeks after the training session, all participants will undergo a different, mannequin-based HFS scenario.

After each simulation, resident performance will be assessed using the Anaesthetists' Non-Technical Skills scale and the Ottawa Crisis Resource Management Global Rating Scale. Evaluators will also perform a summary evaluation with the Managing Emergencies in Pediatric Anesthesia Global Rating Scale.

Resident's satisfaction will be measured with a post-assessment trainee survey scale.

Significance. Should the virtual reality demonstrate to be as efficient as mannequin-based simulation, it will be integrated into the residency curriculum and used for resident training and medical education in institutions that have limited access to a simulation center.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be included if they are residents enrolled in the Anesthesia Residency program at the McGill University

Exclusion Criteria:

* . Participants will be excluded if they refuse or if they have a history of Virtual Reality Induced Symptoms and Effects (VRISE).

Sex: All
Age Groups: Child, Adult, Older Adult